CLINICAL TRIAL: NCT04426097
Title: Effect of Cervical Vagal Blockade on Cough Incidence in Non-intubated Uniportal Video-assisted Thoracoscopic Surgery
Brief Title: Effect of Cervical Vagal Blockade on Cough Incidence in Non-intubated Uniportal Video-assisted Thoracic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TMU-JIRB N201803027
Record Dates: First submitted 2020-03-31; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-03

CONDITIONS: Video-assisted Thoracoscopic Surgery
Keywords: vagus nerve block

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical Vagal Blockade (Experimental)
  Interventions: Procedure: Cervical Vagal Blockade
- Without Blockade (Placebo Comparator)
  Interventions: Procedure: Without Blockade

INTERVENTIONS:
Procedure: Cervical Vagal Blockade — Cervical Vagal Blockade with 0.5 % ropivacaine 2.5 ml and 2% xylocaine 2.5 ml
  Arms: Cervical Vagal Blockade
Procedure: Without Blockade — Without Blockade
  Arms: Without Blockade

SUMMARY:
Currently, there is a trend toward non-intubated anesthesia methods for video-assisted thoracic surgery in our hospital. During the surgery, intrathoracic vagus nerve blockade is suggested for inhibit cough reflex in previous paper. However, right and left side of vagus nerves both deep near the aorta or trachea respectively. To achieving the procedure may induce cough reflex by lobar traction even result vital organ damage. This study aims to apply alternative vagus nerve blockade at neck level via ultrasound guidance and test if the procedure real reduce cough reflex then previous method. We also follow up the patient's vital sign, vocal cord and diaphragm movement, horner syndrome and hoarseness to evaluating if cervical vagal blockade has the potential risk involve other surrounding nerves

ELIGIBILITY:
Inclusion Criteria:

* Adults younger than 80 years old are scheduled for one-port video assisted thoracic surgery

Exclusion Criteria:

* Anticipated difficult airway, Respiratory insufficiency,Vocal cord palsy,diaphragm palsy parkinsonism,previous stroke,tachycardia

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Effect of Cervical Vagal Blockade on Cough Incidence | During the VATS procedure
  number of coughing episodes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katlic MR, Facktor MA. Video-assisted thoracic surgery utilizing local anesthesia and sedation: 384 consecutive cases. Ann Thorac Surg. 2010 Jul;90(1):240-5. doi: 10.1016/j.athoracsur.2010.02.113. PMID 20609784
- [Background] Chen KC, Cheng YJ, Hung MH, Tseng YD, Chen JS. Nonintubated thoracoscopic surgery using regional anesthesia and vagal block and targeted sedation. J Thorac Dis. 2014 Jan;6(1):31-6. doi: 10.3978/j.issn.2072-1439.2014.01.01. PMID 24455173
- [Background] Chen JS, Cheng YJ, Hung MH, Tseng YD, Chen KC, Lee YC. Nonintubated thoracoscopic lobectomy for lung cancer. Ann Surg. 2011 Dec;254(6):1038-43. doi: 10.1097/SLA.0b013e31822ed19b. PMID 21869676
- [Background] Lee YJ, Chung CC, Chou HC, Lin JA. Block for uniportal video-assisted thoracoscopic surgery: an ultrasound-guided, single-penetration, double-injection approach. Br J Anaesth. 2015 Nov;115(5):792-4. doi: 10.1093/bja/aev327. No abstract available. PMID 26475808
- [Background] Dong Q, Liang L, Li Y, Liu J, Yin W, Chen H, Xu X, Shao W, He J. Anesthesia with nontracheal intubation in thoracic surgery. J Thorac Dis. 2012 Apr 1;4(2):126-30. doi: 10.3978/j.issn.2072-1439.2012.03.10. PMID 22833817
- [Background] Giovagnorio F, Martinoli C. Sonography of the cervical vagus nerve: normal appearance and abnormal findings. AJR Am J Roentgenol. 2001 Mar;176(3):745-9. doi: 10.2214/ajr.176.3.1760745. PMID 11222217
- [Background] Arsanious D, Khoury S, Martinez E, Nawras A, Filatoff G, Ajabnoor H, Darr U, Atallah J. Ultrasound-Guided Phrenic Nerve Block for Intractable Hiccups following Placement of Esophageal Stent for Esophageal Squamous Cell Carcinoma. Pain Physician. 2016 May;19(4):E653-6. PMID 27228533
- [Background] Elias M. Cervical sympathetic and stellate ganglion blocks. Pain Physician. 2000 Jul;3(3):294-304. PMID 16906187
- [Background] Polverino M, Polverino F, Fasolino M, Ando F, Alfieri A, De Blasio F. Anatomy and neuro-pathophysiology of the cough reflex arc. Multidiscip Respir Med. 2012 Jun 18;7(1):5. doi: 10.1186/2049-6958-7-5. PMID 22958367